CLINICAL TRIAL: NCT03718052
Title: Early Valve Surgery Versus Conventional Treatment in Infective Endocarditis Patients With High Risk of Embolism: a Randomized Superiority Clinical Trial
Brief Title: Early Valve Surgery Versus Conventional Treatment in Infective Endocarditis Patients With High Risk of Embolism
Acronym: CHIRURGENDO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P160952J
Record Dates: First submitted 2018-10-10; First posted 2018-10-24 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Endocarditis
MeSH Terms: conditions — Endocarditis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early valve surgery (EVS) (Experimental): Cardiac surgery as soon as possible within 72 hours of randomization
  Interventions: Procedure: Early valve surgery (EVS)
- Conventional care (Active Comparator): Conventional care according to the 2015 European guidelines.
  Interventions: Procedure: Conventional Care

INTERVENTIONS:
Procedure: Early valve surgery (EVS) — Early valve surgery (EVS) within 72 hours of randomization
  Arms: Early valve surgery (EVS)
Procedure: Conventional Care — Conventional care according to the 2015 European guidelines.
  Arms: Conventional care

SUMMARY:
Infective endocarditis (IE) is associated with an overall in-hospital mortality rate of 15-25% and a high incidence of embolic events (20-50%). Leading causes of mortality are heart failure (HF) resulting from valve dysfunction, and stroke caused by vegetation embolization. The rate of symptomatic embolic events occurring after antibiotic initiation is around 15%. Valve surgery benefit has been clearly demonstrated in patients with periannular complications and moderate to severe HF resulting from acute valve regurgitation. The timing of surgery to prevent embolism is critical since the risk of new embolic event is highest during the first weeks of antibiotic treatment.

The primary objective is to compare clinical outcomes of Early Valve Surgery (as soon as possible within 72 hours of randomization) with those of a conventional management based on current guidelines in patients with native left-sided IE and high risk of embolism.

208 patients (104 patients per arm) will be included in a national multicenter (21 centers) prospective randomized open blinded end-point (PROBE) sequential superiority trial.

DETAILED DESCRIPTION:
Infective endocarditis (IE) is associated with an overall in-hospital mortality rate of 15-25% and a high incidence of embolic events (20-50%). Leading causes of mortality are heart failure (HF) resulting from valve dysfunction, and stroke caused by vegetation embolization. The rate of symptomatic embolic events occurring after antibiotic initiation is around 15%. Valve surgery benefit has been clearly demonstrated in patients with periannular complications and moderate to severe HF resulting from acute valve regurgitation. Indications of valve surgery for prevention of embolic complications are less clearly defined. Potential complications of valve surgery and of implanted permanent prosthetic valve are to be balanced against their potential benefits in terms of prevented embolism and improved survival. The timing of surgery to prevent embolism is critical since the risk of new embolic event is highest during the first weeks of antibiotic treatment. The points in favor of early valve surgery (EVS) in patients with high embolic risk include the following 1) patients with high risk of embolism are identified by transesophageal echocardiography (TOE); 2) advances in surgical management of IE dramatically lowered postoperative mortality; 3) 2015 European ESC IE guidelines state that valve surgery should be performed in IE with vegetation above 10 mm AND an embolic event occurring while patients are receiving antibiotic (grade I/B) and should be considered in IE with vegetation above 30 mm (Grade IIaB ) and may be above 10 mm and severe valve regurgitation.

The primary objective is to compare clinical outcomes of EVS (as soon as possible within 72 hours of randomization) with those of a conventional management based on current 2015 European ESC guidelines in patients with native left-sided IE and high risk of embolism.

The primary assessment criterion is a composite of all-cause death and clinically symptomatic embolic events within 6 weeks from randomization in all included patient.

208 patients (104 patients per arm) will be included in a national multicenter (21 centers) prospective randomized open blinded end-point (PROBE) sequential superiority trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Definite or possible IE based on the modified Duke criteria (ESC 2015)
3. Length of vegetation on native aortic and/or mitral valve, as assessed by TOE * :

   * between 10 and 15 mm AND (severe regurgitation OR previous symptomatic or asymptomatic embolic events)
   * OR above or equal to 15 mm
4. Initiation of specific IE active antibiotic less than 5 days (≤120 hours) before inclusion
5. For non-menopause women: negative blood or urinary β-HCG test. *If the patient has several vegetations, only one vegetation with these criterions, is enough to included patient.

Exclusion Criteria:

1. Patient with "emergent" indication of surgery based on 2015 European Guidelines
2. Prosthetic valve endocarditis
3. Patient who is not candidate for surgery due to high risk post-surgery mortality including for example coexisting major embolic stroke with a high risk of hemorrhagic transformation, symptomatic hemorrhagic stroke; poor medical status, such as coexisting malignancies…
4. No written informed consent from the patient or a legal representative if appropriate
5. Patient with no national health or universal plan affiliation coverage
6. Pregnancy
7. Patient under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Complications and deaths in all included patient | Week 6
  A composite of all-cause death and clinically symptomatic embolic events within 6 weeks from randomization in all included patient.

SECONDARY OUTCOMES:
Complications and deaths in patient with definite IE | Week 6
  All-cause death and clinically symptomatic embolic events from randomization in patient with definite IE
Complications and deaths | Months 6 and 12
  Combination of all-cause death and clinically symptomatic embolic events documented by imaging studies up to 6 months and one-year after randomization.
Deaths | Months 6 and 12
  All-cause death up to 6 months and one-year (post study analysis) after randomization
Symptomatic embolic events | Months 6 and 12
  All clinically symptomatic embolic events documented by imaging studies up to 6 months and one-year after randomization
Intensive care scale | Week 6 , Months 3, 6 and 12
  Glasgow outcome scale and Rankin scale at week 6, month 3, 6 and one-year visits.
Infective EI relapse | Months 6 and 12
  Relapse of infective IE up to 6 months and one-year after randomization.
Infective EI recurrences | Months 6 and 12
  Recurrences of infective IE up to 6 months and one-year after randomization.
Rehospitalization | Week 6, Months 6 and 12
  Readmission due to development of congestive heart failure up to 6 weeks, 6 months and one-year after randomization
Rehospitalization for valve surgery | Months 6 and 12
  Readmission for valve surgery (between hospital discharge and 6 months and one-year after enrolment) in patients operated on during the acute phase of IE
Thrombosis and ischemia | Months 6 and 12
  Six month and one-year prosthesis thrombosis, severe adverse events due to anticoagulation, ischemic stroke due to documented suboptimal anticoagulation
Quality of life scale 1 | Months 6 and 12
  WhoQol scale up to 6 months and one-year after randomization.
Quality of life scale 2 | Months 6 and 12
  SF36 up to 6 months and one-year after randomization.
Delay between randomization and surgery | Months 12
  Time interval between randomization and date of cardiac surgery in patients operated-on during the acute phase of the IE.

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Duval, Principal Investigator — Bichat Hospital
Locations (1):
- Bichat Claude Bernard Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided